CLINICAL TRIAL: NCT06991777
Title: Feasibility Study: Precision Sedation in Intensive Care Using Neurophysiologic and Respiratory Targets.
Brief Title: Precision Sedation in Intensive Care
Acronym: SENSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Theresa Mariero Olasveengen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-04923
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness
Keywords: sedation; critical care; EEG; neurophysiology; respiratory
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Precision sedation in intensive care using neurophysiologic and respiratory targets. (Experimental): Precision sedation in intensive care using neurophysiologic and respiratory targets.
  Interventions: Device: Precision sedation in intensive care using neurophysiologic and respiratory targets.
- Control (No Intervention): Sedation titration using standardized assessments (Richmond Agitation-Sedation Scale (RASS))

INTERVENTIONS:
Device: Precision sedation in intensive care using neurophysiologic and respiratory targets. — Sedation titration using EEG and ventilator parameters
  Arms: Precision sedation in intensive care using neurophysiologic and respiratory targets.

SUMMARY:
Being critically ill and in need of mechanical ventilation is painful and distressing, and patients rarely have the capacity to communicate to express their needs. Doctors and nurses caring for critically ill patients in need of mechanical ventilation are constantly trying to balance patient comfort vs. patient safety. On one hand health care personnel (HCP) want to avoid unnecessary pain and suffering, on the other hand HCP want our patients to be able to communicate and avoid the complications associated with prolonged mechanical ventilation and Intensive Care Unit (ICU) stays. Our current tools for titrating sedation are subjective and variable, leading to large variations in sedation strategy between providers and frequent oversedation to "err on the side of caution".

This project is a grassroot initiative where physicians and nurses across various ICUs at Oslo University Hospital are highly motivated to research an alternative strategy for sedation in our units. The investigators believe a more precise approach to sedation that uses neurophysiologic and respiratory targets to guide medication dosing will significantly improve our overall quality of care. By avoiding oversedation, the investigators hope to help our patients wean off mechanical ventilation quicker, reduce their risk of delirium and cognitive deficit, resulting in fewer complications and shorter ICU stays. More precise sedation not only has the potential to improve outcomes for individual patients, but it can also improve ICU capacity and reduce the costs associated with prolonged ICU stays.

DETAILED DESCRIPTION:
1. INTRODUCTION A significant proportion of the patients admitted to an intensive care unit (ICU) undergo mechanical ventilation.1,2 It is common practice to administer sedative and analgesic drugs to these patients, to improve their comfort and their interaction with the ventilator. Careful titration of analgesia and sedation is important to prevent pain and discomfort in this population of patients, but oversedation has been associated with increased mortality and morbidity. Optimizing sedation practice may reduce mortality, duration of mechanical ventilation and ICU length of stay, resulting in reduced costs and improved resource utilization. The recommended strategy is to titrate sedation using scales or scores based on clinical criteria.6 There is variability in the specific domains they assess (e.g. consciousness, cognition, and comprehension), and in their implementation (about 88% of units use a sedation scale, with variability in the sedation scale used). There is also an inherent subjectiveness to these scales, with important variability among healthcare providers resulting in significant over-sedation in the ICU.

   The current Pain, Agitation/sedation, Delirium, Immobility and Sleep disruption (PADIS) guidelines focuses on early rehabilitation and quick ventilator liberation, but has become criticized for relying on clinical sedation scores to guide sedation alone. A panel of experts, mostly from the collaborative group who authored the PADIS guidelines, have recently provided an updated "state of the art" narrative review to support clinicians in their management of sedation/analgesia with a revised "ABCDEF-R" bundle (R = Respiratory-drive control). This review highlights giving priority to the management of mechanical-ventilator and respiratory-drive related factors to avoid the unnecessary use of medications. As arousal level poorly correlates with markers of patient respiratory effort, and some potentially injurious ventilator dyssynchrony may actually be exacerbated by deeper sedation15 there is a need for new sedation titration strategies less reliant on scales that only assess arousal.

   New techniques and devices (such as Bispectral Index, State Entropy, Auditory evoked potentials, Narcotrend Index, Patient State Index monitoring) have been developed with the purpose of providing an objective measurement of patient's sedation. The Bispectral Index monitor is possibly the most studied and adapted. Bispectral Index monitoring is based on the processing of electroencephalographic signals from the brain. The device uses three or four electrodes applied to the patient's forehead. The electrodes record the raw frontal electroencephalogram (EEG) signal and process it through both standard and proprietary algorithms to provide processed EEG parameters of brain electrical activity. These parameters correlate to various states of wakefulness, and can also measure and quantify burst suppression, a specific pattern of brain activity that indicates deep coma with severely reduced brain activity. Although induction of burst suppression using sedatives can be warranted in special circumstances such as status epilepticus, it is normally considered a measurement of over-sedation.

   Bispectral Index or EEG monitoring is quite well established for monitoring anaesthesia depth. Recent studies have shown that titrating anaesthesia depth towards a goal of a Bispectral Index between 50-60 and avoiding burst suppression yields less delirium, shorter stay in recovery and for certain vulnerable groups improved cognitive function when tested 1 year after anesthesia. The usefulness of Bispectral Index or EEG monitoring in the ICU setting has been considerably less studied. A recent Cochrane systematic review only identified four studies (256 participants) comparing processed EEG guided sedation to standard care. These studies had severe limitations; one study (50 adults) failed to demonstrate reduced length of ICU stay, two studies (155 adults) failed to demonstrate reduced duration of ventilation, and one study (105 adults) did not find any differences in adverse events. The overall assessment was that the level of evidence is very low, and that there is insufficient evidence to provide any guidance on the use of processed EEG to guide sedation in the ICU.

   This feasibility study is the first step in a larger project to develop and evaluate a novel treatment strategy for sedation during intensive care. The feasibility study seeks to optimize feasibility and safety by identifying optimal inclusion criteria, methods of measuring neurophysiologic and respiratory targets and outcome measures. The results from the pilot study will help guide the final planning and implementation of a larger clinical randomized controlled trial comparing a novel approach to individualized sedation using neurophysiologic and respiratory targets to standard care in multiple intensive care units at Oslo University Hospital.
2. HYPOTHESIS, AIMS AND STUDY OBJECTIVES The planned study will focus on investigating the feasibility and safety of precision sedation in the ICU, using a combination of neurophysiologic and respiratory targets.

   Hypothesis: Precision sedation titrated to neurophysiologic and respiratory targets is safe and feasible.

   Aims and objectives Feasibility Study: Investigate the safety and feasibility of a novel precision sedation strategy.
   1. Compare adverse events such as accidental removal of tubes and lines, use of sedatives, opioids or vasopressors above recommended ranges, or other unexpected adverse events between intervention and control groups.
   2. Evaluate the actual use and perceived clinical usefulness of processed EEG parameters such as Bispectral index, suppression ratio, accumulated suppression time, spectral edge frequency and median frequency, to adjust and improve the sedation titration strategy prior to main trial.
   3. Determine whether length of intensive care stay, time to spontaneous eye opening and time to following commands after daily interruption of sedation, and incidence and duration of delirium are feasible outcomes for a larger clinical trial.
3. PROJECT METHODOLOGY The initial pilot study will evaluate the safety and feasibility of our precision sedation strategy and allow us to refine the neurophysiologic and respiratory elements of the strategy before planning a larger randomized controlled trial. Patients will be randomized to receive either precision sedation or traditional sedation, with dosing guided by clinical assessment alone. The results of these studies have the potential to improve the management of sedation in the ICU, reduce the incidence of adverse outcomes associated with excessive sedation, and improve patient outcomes. The findings will also have important implications for healthcare providers and policymakers, as they may inform the development of guidelines and protocols for sedation management in the ICU.

   3.1 Project arrangements, method selection and analyses The "precision sedation in intensive care" project group is well established and functioning. Infrastructure for continuous patient inclusion and data collection is already in place.

   3.1.1 Study design and statistical power The study is designed as a 100 patient randomized, controlled feasibility trial where 50 patients will be randomized to precision sedation using neurophysiologic and respiratory targets and 50 patients will be randomized to standard care (control group) across three locations - Surgical Intensive Care Units at Oslo University Hospital Ullevål and Rikshospitalet, and Intensive Care Unit, Sorlandet Hospital, Arendal. No formal power analysis is performed for this feasibility study, but 100 patients across two locations should provide enough patients to assess the feasibility of intervention, data collection and analysis for the relevant patient groups.

   3.1.2 Study population Inclusion Criteria 1) All adult (age≥18 years) 2) Admitted to ICU 3) Estimated need for sedation > 24 hours All criteria must be met for inclusion. Exclusion Criteria 1) Patients admitted for palliative care 2) Patients admitted with restrictions in care (no ventilator treatment) 3) Contraindication for daily interruption of sedation Any criteria present leads to exclusion.

   3.1.3 Intervention EEG monitoring will be initiated and recorded for both intervention and control groups immediately after randomization and continue for up to 7 days or until extubation, but health care providers will be blinded for all EEG parameters in the control group.

   3.2 Participants, organization and collaborations The Steering Committee will coordinate the study. Locally, the study will be managed and coordinated by Site Investigators (SI) at each location. The site investigators will be responsible for data collection and maintenance of study documentation.

   3.3 Budget Division of Emergencies and Critical Care, Oslo University Hospital (OUH) is covering costs related to data collection including follow-up, office supplies and some training costs. Costs related to salary for PhD student has been secured from South-Eastern Heath Authority. Costs related to disposable equipment for EEG monitoring has been secured from Charlottefondet.

   3.4 Plan for activities, visibility, and dissemination 2024: Complete data collection, data analysis and interpretation. 2025: Prepare manuscript while using the results from this feasibility study plan for a larger study to evaluate effectiveness of a novel precision sedation strategy.

   3.4 Plan for implementation The results of this study will be highly anticipated within the participating intensive care units. The project will have widespread involvement from health care providers, and the investigators expect the trial results will lead to the planning of a larger randomized controlled trial on precision sedation. The investigators plan to present the feasibility study results at national and international conferences and publish our findings in a peer-reviewed journal.
4. STATISTICAL METHODS AND DATA ANALYSIS The study design is unblinded, but all data analyses will be performed blinded to the allocation to intervention or control to the extent possible. Data will be analysed by the intention-to-treat principle. Continuous data will be presented as mean ± standard deviation (SD) or median (quartiles) depending on data distribution. Categorical data will be presented as number of total (%). Continuous efficacy variables will be analysed using independent T-tests for comparisons between the treatment arms. Categorical data will be compared using Chi-square with continuity correction. If necessary, values will be log-transformed to meet the assumptions of the tests. Temporal trends between groups will be compared using a generalised mixed model with an unstructured covariance matrix.
5. USER INVOLVEMENT The investigators plan to recruit a user representative to the steering committee to ensure user involvement in the practical planning of the study. The study will be presented for and discussed with the research committee at the Division of Emergencies and Critical Care, Oslo University Hospital. The research committee is multidisciplinary with user representation, and their insights and suggestions will be sought throughout the planning, execution and dissemination phase of this study. Ethical aspects of conducting research on unconscious patients unable to consent prior to inclusion will be discussed specifically.
6. ETHICAL CONSIDERATIONS This study will be conducted according to the principles of the Declaration of Helsinki as stated in the current version of Fortaleza, Brazil, 2013. The protocol and any subsequent modifications will be reviewed and approved by the Regional Ethical Committee South-East, and Data Protection Officer, Oslo University Hospital.

Whenever possible, informed written consent will be obtained prior to study inclusion. For patients unable to provide informed consent at time of randomization the investigators will seek advice from the regional ethics committee and the Oslo University Hospital Data Protection Officer. In previous studies including patients unable to provide consent the regional ethics committee has advised including and randomizing without consent based on family consultation. Final written consent has then been obtained as soon as the patients was deemed able to provide informed consent. The investigators will adhere to the procedures mandated by the regional ethics committee and Data Protection Officer. Patient autonomy to withdraw from the study at any time will be respected.

All participating researchers are obliged to declare any conflicts of interest or financial interest related to the study.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU
* Estimated need for sedation > 24 hours

Exclusion Criteria:

* Patients admitted for palliative care
* Patients admitted with restrictions in care (no ventilator treatment)
* Contraindication for daily interruption of sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Completeness of data in CRF | through study completion, an average of 7 days
  Evaluate feasibility of recording all available processed EEG parameters (Bispectral index, suppression ratio, accumulated suppression time, spectral edge frequency and median frequency) and report as percentage of missing values. This information is to be used to adjust and improve data capture strategy prior to main trial.

SECONDARY OUTCOMES:
Reported Adverse events (Safety) | through study completion, an average of 7 days
  Compare adverse events such as accidental removal of tubes and lines, use of sedatives, opioids or vasopressors above recommended ranges, or other unexpected adverse events between intervention and control groups.
Length of intensive care stay | through study completion, an average of 7 days
  Determine whether length of intensive care stay (number of days) is a feasible outcome for a larger clinical trial.
Time to spontaneous eye opening | through study completion, an average of 7 days
  Determine whether time to spontaneous eye opening (number of days) is a feasible outcome for a larger clinical trial.
Time to following commands | through study completion, an average of 7 days
  Determine whether time to following commands (number of days) is a feasible outcome for a larger clinical trial.
Incidence of delirium | through study completion, an average of 7 days
  Determine whether incidence of delirium (number with delirium in treatment and control group) is a feasible outcome for a larger clinical trial.
Duration of delirium | through study completion, an average of 7 days
  Determine whether duration of delirium (number of days) is a feasible outcome for a larger clinical trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because this is a pilot study with a small sample size, limiting the generalisability and reusability of the data. Additionally, participants did not provide specific consent for data sharing, and institutional policies restrict dissemination of individual-level data. The study also lacks the resources and infrastructure needed for secure data curation and anonymisation.

REFERENCES:
- [Background] Zhao D, Xu Y, He W, Li T, He Y. [A comparison of bispectral index and sedation agitation scale in guiding sedation therapy: a randomized controlled study in patients undergoing short term mechanical ventilation]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2011 Apr;23(4):220-3. Chinese. PMID 21473824
- [Background] Weatherburn C, Endacott R, Tynan P, Bailey M. The impact of bispectral index monitoring on sedation administration in mechanically ventilated patients. Anaesth Intensive Care. 2007 Apr;35(2):204-8. doi: 10.1177/0310057X0703500208. PMID 17444309
- [Background] Rasulo FA, Hopkins P, Lobo FA, Pandin P, Matta B, Carozzi C, Romagnoli S, Absalom A, Badenes R, Bleck T, Caricato A, Claassen J, Denault A, Honorato C, Motta S, Meyfroidt G, Radtke FM, Ricci Z, Robba C, Taccone FS, Vespa P, Nardiello I, Lamperti M. Processed Electroencephalogram-Based Monitoring to Guide Sedation in Critically Ill Adult Patients: Recommendations from an International Expert Panel-Based Consensus. Neurocrit Care. 2023 Apr;38(2):296-311. doi: 10.1007/s12028-022-01565-5. Epub 2022 Jul 27. PMID 35896766
- [Background] Punjasawadwong Y, Phongchiewboon A, Bunchungmongkol N. Bispectral index for improving anaesthetic delivery and postoperative recovery. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD003843. doi: 10.1002/14651858.CD003843.pub3. PMID 24937564
- [Background] Carrasco G. Instruments for monitoring intensive care unit sedation. Crit Care. 2000;4(4):217-25. doi: 10.1186/cc697. Epub 2000 Jul 13. PMID 11094504
- [Background] Akoumianaki E, Lyazidi A, Rey N, Matamis D, Perez-Martinez N, Giraud R, Mancebo J, Brochard L, Richard JM. Mechanical ventilation-induced reverse-triggered breaths: a frequently unrecognized form of neuromechanical coupling. Chest. 2013 Apr;143(4):927-938. doi: 10.1378/chest.12-1817. PMID 23187649
- [Background] Dzierba AL, Khalil AM, Derry KL, Madahar P, Beitler JR. Discordance Between Respiratory Drive and Sedation Depth in Critically Ill Patients Receiving Mechanical Ventilation. Crit Care Med. 2021 Dec 1;49(12):2090-2101. doi: 10.1097/CCM.0000000000005113. PMID 34115638
- [Background] Chanques G, Constantin JM, Devlin JW, Ely EW, Fraser GL, Gelinas C, Girard TD, Guerin C, Jabaudon M, Jaber S, Mehta S, Langer T, Murray MJ, Pandharipande P, Patel B, Payen JF, Puntillo K, Rochwerg B, Shehabi Y, Strom T, Olsen HT, Kress JP. Analgesia and sedation in patients with ARDS. Intensive Care Med. 2020 Dec;46(12):2342-2356. doi: 10.1007/s00134-020-06307-9. Epub 2020 Nov 10. PMID 33170331
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Quigley F, Rosenberg JM, Shachar-Hill Y, Bohnert HJ. From genome to function: the Arabidopsis aquaporins. Genome Biol. 2002;3(1):RESEARCH0001. doi: 10.1186/gb-2001-3-1-research0001. Epub 2001 Dec 7. PMID 11806824
- [Background] Soliman HM, Melot C, Vincent JL. Sedative and analgesic practice in the intensive care unit: the results of a European survey. Br J Anaesth. 2001 Aug;87(2):186-92. doi: 10.1093/bja/87.2.186. PMID 11493487
- [Background] Martin J, Franck M, Sigel S, Weiss M, Spies C. Changes in sedation management in German intensive care units between 2002 and 2006: a national follow-up survey. Crit Care. 2007;11(6):R124. doi: 10.1186/cc6189. PMID 18062820
- [Background] Reschreiter H, Maiden M, Kapila A. Sedation practice in the intensive care unit: a UK national survey. Crit Care. 2008;12(6):R152. doi: 10.1186/cc7141. Epub 2008 Dec 1. PMID 19046459
- [Background] Sessler CN, Varney K. Patient-focused sedation and analgesia in the ICU. Chest. 2008 Feb;133(2):552-65. doi: 10.1378/chest.07-2026. PMID 18252923
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253
- [Background] Jackson DL, Proudfoot CW, Cann KF, Walsh T. A systematic review of the impact of sedation practice in the ICU on resource use, costs and patient safety. Crit Care. 2010;14(2):R59. doi: 10.1186/cc8956. Epub 2010 Apr 9. PMID 20380720
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Background] Kollef MH, Levy NT, Ahrens TS, Schaiff R, Prentice D, Sherman G. The use of continuous i.v. sedation is associated with prolongation of mechanical ventilation. Chest. 1998 Aug;114(2):541-8. doi: 10.1378/chest.114.2.541. PMID 9726743
- [Background] Metnitz PG, Metnitz B, Moreno RP, Bauer P, Del Sorbo L, Hoermann C, de Carvalho SA, Ranieri VM; SAPS 3 Investigators. Epidemiology of mechanical ventilation: analysis of the SAPS 3 database. Intensive Care Med. 2009 May;35(5):816-25. doi: 10.1007/s00134-009-1449-9. Epub 2009 Mar 14. PMID 19288079
- [Background] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214